CLINICAL TRIAL: NCT05132621
Title: The Genital Tract Microflora in Women With Systemic Lupus Erythematosus and IgA Nephropathy.
Brief Title: The Genital Tract Microflora in Women With Systemic Lupus Erythematosus (SLE) and Immunoglobulin A (IgA) Nephropathy.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: SLEIGA-1
Record Dates: First submitted 2021-11-22; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Systemic Lupus Erythematosus; Immunoglobulin A Nephropathy
Keywords: microbiome; systemic lupus erythematosus; IgA nephropathy
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Vaginal secretion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants diagnosed with SLE
  Interventions: Diagnostic Test: Smear
- Participants diagnosed with IgA nephropathy
  Interventions: Diagnostic Test: Smear
- Healthy Participants
  Interventions: Diagnostic Test: Smear

INTERVENTIONS:
Diagnostic Test: Smear — A smear of the posterior vaginal fornix collected with a gynecological speculum.

SUMMARY:
The study hypothesis:

Systemic lupus erythematosus (SLE) is a chronic autoimmune disease with a broad spectrum of clinical manifestations. Its mechanisms are not well understood. It is known that its development is influenced by genetic factors and gender. However, it is believed that in some patients with a specific genetic predisposition, certain environmental factors such as chemicals, including drugs and toxins, smoking, or infections may initiate the development of the disease. Of particular importance seem to be infections, which by stimulating the immune system can induce new symptoms or exacerbate existing ones.

For this reason, links between the microbiome and the clinical course of SLE are being sought. Most available studies concern the intestinal microbiome. So far, the relationship between the genital tract microbiota and the clinical picture of SLE has not been documented.

Aim of the study:

This study aims to identify and differentiate the genital tract microbiota of women with a diagnosis of systemic lupus, IgA nephropathy and a control group of healthy women. The results will be correlated with the clinical presentation of these diseases. In addition, the isolated bacterial strains will be secured for further study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years,
* Confirmed diagnosis of SLE or IgA nephropathy,
* First half of the menstrual cycle, after the end of bleeding,
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Lack of menstruation,
* Pregnancy,
* Active infection requiring parenteral or topical antibiotic therapy within 2 weeks before examination,
* Neoplastic disease of the reproductive tract.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — A study based on the analysis of genital tract microflora of women of reproductive age.
Study Population: 50 participants diagnosed with SLE and 50 participants diagnosed with IgA nephropathy will be included in the study. The control group will consist of 50 healthy participants.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Differences in microflora composition between groups of study participants | Two months

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Immunology, Transplantology and Internal Medicine Transplantation Institute, Warsaw Medical University, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided